CLINICAL TRIAL: NCT05021263
Title: Does IV Magnesium Improve Quality of Recovery With ERAS Protocols in Laparoscopic Colorectal Surgery?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Kevin Min, Assistant Professor, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21D.499
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Colo-rectal Cancer; Anesthesia
MeSH Terms: conditions — Colonic Neoplasms | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Magnesium Group (Experimental): The magnesium group (Mg) will receive a bolus of 50 mg/kg of IV magnesium prior to incision and an infusion of 15 mg/kg/hr, with no preoperative oral pregabalin. All groups will receive preoperative oral acetaminophen, preoperative NSAIDs, subcutaneous heparin, intraoperative TAP block, intraoperative dexamethasone, ondansetron, transdermal scopolamine patch, and postoperative care as per the current ERAS protocol.
  Interventions: Drug: IV Medications
- Control Group (Placebo Comparator): The control group (Ct) will receive saline solution and no IV magnesium or oral pregabalin. All groups will receive preoperative oral acetaminophen, preoperative NSAIDs, subcutaneous heparin, intraoperative TAP block, intraoperative dexamethasone, ondansetron, transdermal scopolamine patch, and postoperative care as per the current ERAS protocol.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: IV Medications — IV magnesium sulfate, used to replete magnesium stores
  Arms: Magnesium Group
Other: placebo — placebo
  Arms: Control Group

SUMMARY:
This study is a randomized, double blind controlled trial examining the impact of incorporating a single intraoperative intravenous magnesium bolus and infusion into a preexisting Enhanced Recovery After Surgery (ERAS) protocol for colorectal surgery in place of preoperative oral pregabalin. These protocols are pathways designed with the goal of achieving early surgical recovery by utilizing a constellation of perioperative care techniques that include the use of opioid-sparing pain medications, minimally invasive approaches, and prevention of post-operative nausea and vomiting, among others. Intravenous magnesium has shown to be an effective non-opioid analgesic in abdominal surgeries that decreases total opioid consumption, pain, and improves recovery. The purpose of this study is to evaluate whether or not the addition of intravenous magnesium to our institutional ERAS protocol will improve specific outcome measures, and provide additional benefits when compared to oral preoperative pregabalin. The primary outcome is the patient's quality of recovery based on the "Quality of Recovery - 40 Questionnaire" (QOR 40), and secondary outcomes will be opioid consumption, pain, shivering, sedation scores, acute kidney injury, gastrointestinal function, respiratory function, and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Elective Laparoscopic Colorectal Surgery
* Age 18-75
* ASA (American Society of Anesthesiologists) Physical Status Classification 1-3

Exclusion Criteria:

* Current use of Buprenorphine/Suboxone or Methadone maintenance treatment
* Known history of substance abuse
* Use of intra- and/or postoperative Ketamine or Lidocaine infusion
* Pre- or postoperative placement of Epidural catheter
* Inability to speak English or communicate verbally
* Chronic Kidney Disease (CKD) Stage 3
* Hepatic Cirrhosis
* Neuromuscular disease
* Heart block on EKG
* Uncontrolled diabetes with Hba1c > 8%
* Known allergies to study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 40 Questionnaire | Postoperative Day 0-2
  Validated Assessment of Postoperative Recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided